CLINICAL TRIAL: NCT07260812
Title: A Phase I Clinical Study on the Safety, Tolerability, and Efficacy of KSV01 Injection in Patients With Relapsed/Refractory B-Cell Non-Hodgkin Lymphoma
Brief Title: KSV01 Injection for the Treatment of Relapsed/Refractory B-cell Non-Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: TCRx Therapeutics Co.Ltd (Industry)
Collaborators: Tongji Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSV01-R101
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KSV01 Injection (Experimental): KSV01 Injection is one kind of third-generation non-replicative self-inactivating lentivirus vector which carries CD19 CAR.
  Interventions: Drug: KSV01 Injection

INTERVENTIONS:
Drug: KSV01 Injection — KSV01 Injection is one kind of third-generation non-replicative self-inactivating lentivirus vector which carries CD19 CAR.

SUMMARY:
This is a single center, single arm, open-label, dose escalation, phase 1 study to evaluate the safety, tolerability and preliminary efficacy of KSV01 Injection for patients with B-cell non-hodgkin lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients or their legal guardians voluntarily participate in the study and provide written informed consent.
2. Aged 18 to 80 years (inclusive), male or female.
3. ECOG performance status score of ≤ 1.
4. Life expectancy > 3 months.
5. KPS score ≥ 70.
6. Patients with B-cell non-Hodgkin lymphoma (B-NHL) diagnosed according to the 2016 WHO classification, with priority given to the following pathological types: DLBCL (NOS; including DLBCL transformed from indolent NHL), PMBCL, FL3b, and HGBCL (including double-hit/triple-hit lymphomas).
7. CD19 positivity confirmed by flow cytometry and/or histopathology (Documented prior CD19 positivity confirmed by the investigator is acceptable). Subjects who have received prior anti-CD19 therapy must undergo a biopsy to confirm current CD19 positive expression.
8. According to the Lugano 2014 criteria, the presence of PET-positive target lesions for tumor assessment is required (Deauville 5-Point Scale [5-PS] ≥ 4).
9. Adequate organ function:

   1. Hepatic function: ALT ≤ 5 times the upper limit of normal (ULN) and total bilirubin < 2.0 mg/dL (< 3.0 mg/dL for patients with Gilbert's syndrome or documented lymphomatous infiltration of the liver);
   2. Renal function: Creatinine clearance (calculated by Cockcroft-Gault formula) ≥ 60 mL/min;
   3. Pulmonary function: Oxygen saturation (SaO₂) ≥ 92% on room air, and no active pulmonary infection;
   4. Cardiac function: Left ventricular ejection fraction (LVEF) ≥ 40% by echocardiography, absence of significant pericardial effusion, and no clinically significant electrocardiogram (ECG) abnormalities.
10. Female patients of childbearing potential must have a negative urine/blood pregnancy test during the screening period and agree to use effective contraception for at least 1 year after infusion; male subjects with partners of childbearing potential must agree to use effective barrier contraception for at least 1 year after infusion.

Exclusion Criteria:

1. History of another primary malignancy that has not been in continuous remission for at least 2 years, except for the following conditions which are exempt from the 2-year limit: non-melanoma skin cancer, Stage I solid tumors treated with curative intent and low risk of recurrence, cured localized prostate cancer, biopsy-confirmed carcinoma in situ of the cervix, or squamous intraepithelial lesion identified on Pap smear.
2. Uncontrolled infectious disease within 4 weeks prior to enrollment.
3. Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
4. HIV infection.
5. Positive for Treponema pallidum(syphilis).
6. Severe autoimmune disease or immunodeficiency, with the exception of well-controlled Type I diabetes and thyroid disorders.
7. History of severe allergy or hypersensitivity to macromolecular biologic agents (e.g., antibodies, cytokines).
8. Participation in any other clinical trial within 4 weeks prior to enrollment.
9. History of clinically significant central nervous system (CNS) diseases, including but not limited to epilepsy, paresis, aphasia, stroke, severe head injury, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome.
10. Presence of isolated CNS involvement by lymphoma, or any ongoing CNS condition that precludes accurate neurological evaluation.
11. History of any of the following cardiovascular conditions within the past 6 months: Class III or IV heart failure as defined by the New York Heart Association (NYHA), cardiac angioplasty or stenting, myocardial infarction, unstable angina, or other clinically significant heart disease.
12. Presence of psychiatric illness.
13. History of drug abuse or addiction.
14. Use of the following medications or therapies:

    1. Corticosteroids: Therapeutic doses of corticosteroids (defined as prednisone or equivalent >20 mg/day) within 72 hours prior to study drug infusion; physiologic replacement doses, and topical or inhaled steroids are permitted.
    2. Chemotherapy: Salvage chemotherapy within 2 weeks prior to study drug infusion.
    3. GvHD Therapy: Anti-graft-versus-host disease (GvHD) therapy within 4 weeks prior to study drug infusion.
    4. Allogeneic hematopoietic stem cell transplantation.
    5. Gene therapy.
    6. Adoptive cell therapy.
    7. Prior treatment with alemtuzumab within 6 months, or cladribine or clofarabine within 3 months prior to study drug infusion.
    8. Radiotherapy: Radiotherapy within 6 weeks prior to signing informed consent. To be eligible, lesions within the radiation field must have shown disease progression (PD), or the patient must have PET-positive lesions outside the radiation field. If PET-positive lesions exist outside the radiation field, radiotherapy to other lesions must have been completed at least 2 weeks prior to the first study drug dose.
15. Women who are breastfeeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting Toxicity | 28 days after administration
  DLT evaluation period: The DLT evaluation period is defined as within 28 days (inclusive) after the subjects' first administration of KSV01 injection during the dose escalation stage. All adverse events should be graded and evaluated in accordance with CTCAE v5.0. Among them, cytokine release syndrome (CRS) and immune effector cell-related neurotoxicity syndrome (ICANS) should be determined and graded in accordance with the standards of the American Society for Transplantation and Cell Therapy (ASTCT).

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No